CLINICAL TRIAL: NCT02805725
Title: Targeting Microenvironment and Cellular Immunity in Sarcomas Weekly Trabectedin Combined With Metronomic Cyclophosphamide (CP) in Patients With Advanced Pretreated Soft-tissue Sarcomas. A Phase I/II Study From the French Sarcoma Group.
Brief Title: Targeting Microenvironment and Cellular Immunity in Sarcomas Weekly Trabectedin Combined With Metronomic Cyclophosphamide
Acronym: TARMIC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB 2015-04
Record Dates: First submitted 2016-05-25; First posted 2016-06-20 (Estimated); Results first posted 2023-03-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Soft-tissue Sarcomas
Keywords: Advanced solid tumor; Advanced pretreated soft tissue sarcomas; Phase I/II trial; Dose escalation; PK study
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: Trabectedin 0.30 mg/m2 IV + CP (Experimental): Trabectedin 0.30 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 1 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Interventions: Drug: Phase 1: Trabectedin; Drug: Phase 1: Cyclophosphamide
- Cohort 2: Trabectedin 0.40 mg/m2 IV + CP (Experimental): Trabectedin 0.40 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 2 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Interventions: Drug: Phase 1: Trabectedin; Drug: Phase 1: Cyclophosphamide
- Cohort 3: Trabectedin 0.50 mg/m2 IV + CP (Experimental): Trabectedin 0.50 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 3 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Interventions: Drug: Phase 1: Trabectedin; Drug: Phase 1: Cyclophosphamide
- Cohort 4: Trabectedin 0.60 mg/m2 IV + CP (Experimental): Trabectedin 0.60 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 4 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Interventions: Drug: Phase 1: Trabectedin; Drug: Phase 1: Cyclophosphamide
- Phase II: Trabectedin 0.50 mg/m2 IV + CP (Experimental): Trabectedin 0.50 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in the phase II part of the study.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Interventions: Drug: Phase 2: Trabectedin; Drug: Phase 2: Cyclophosphamide

INTERVENTIONS:
Drug: Phase 1: Trabectedin — Phase I trial based on a dose escalating study design (3+3 traditional design) assessing four dose levels of Trabectedin in combination with metronomic cyclophosphamide (CP).
  A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.)
  Arms: Cohort 1: Trabectedin 0.30 mg/m2 IV + CP; Cohort 2: Trabectedin 0.40 mg/m2 IV + CP; Cohort 3: Trabectedin 0.50 mg/m2 IV + CP; Cohort 4: Trabectedin 0.60 mg/m2 IV + CP
Drug: Phase 2: Trabectedin — Patients will be included in a single-arm phase II trial. Administrated dose will be the RP2D defined in the dose escalation part of the trial. The design will follow a two-stage Simon's optimal design.
  All patients will be treated at the RP2D of trabectedin defined in the preliminary phase I trial with the same schedule as in the phase I trial.
  Arms: Phase II: Trabectedin 0.50 mg/m2 IV + CP
Drug: Phase 1: Cyclophosphamide — A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  Arms: Cohort 1: Trabectedin 0.30 mg/m2 IV + CP; Cohort 2: Trabectedin 0.40 mg/m2 IV + CP; Cohort 3: Trabectedin 0.50 mg/m2 IV + CP; Cohort 4: Trabectedin 0.60 mg/m2 IV + CP
Drug: Phase 2: Cyclophosphamide — All patients will be treated with metronomic cyclophosphamide with the same schedule as in the phase I trial.
  Arms: Phase II: Trabectedin 0.50 mg/m2 IV + CP

SUMMARY:
Assessment of the efficacy and safety of trabectedin and metronomic cyclophosphamide (CP) in patients with advanced pretreated soft-tissue sarcomas, once the Maximum Tolerated Dose (MTD) have been determined (phase I trial).

DETAILED DESCRIPTION:
Phase I: Multicenter Phase I trial based on a dose escalation study design (3+3 traditional design). Phase II: One-arm, multicenter Phase II trial based on two-stage optimal Simon's design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with soft-tissue sarcoma histologically confirmed by central review
2. Metastatic or unresectable locally advanced disease,
3. Age ≥ 18 years,
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2,
5. Life expectancy > 3 months,
6. Measurable disease according to RECIST v1.1 outside any previously irradiated field,
7. For patients included in phase II study, progressive disease according to RECIST v1.1 criteria diagnosed on the basis of two CT scan or MRI obtained at an interval less than 6 months in the period of 12 months prior to inclusion and confirmed by central review,
8. Previous use of Anthracyclines,
9. Have provided tissue from an archival tissue sample,
10. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy,
11. Adequate hematological, renal, metabolic and hepatic function:

    1. Hemoglobin ≥ 9 g/dl (patients may have received prior red blood cell [RBC] transfusion, if clinically indicated); absolute neutrophil count (ANC) ≥ 1.5 x 10^9/l, and platelet count ≥ 100 x 10^9/l
    2. Alanine aminotransferase (ALT), aspartate aminotransferase (AST)< or = 2.5 x upper limit of normality (ULN) ( < or = 5 in case of extensive liver involvement) and alkaline phosphatase (AP) < or = 2.5 x ULN
    3. Total bilirubin < or = ULN.
    4. Albumin ≥ 25 g/l
    5. Serum Creatinine < or =1.5 x ULN or calculated creatinine clearance (CrCl) ≥ 30 ml/min (according to Cockroft formula).
    6. Creatine Phosphokinase (CPK) < or = 2.5 x ULN
12. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for six months after discontinuation of treatment. Acceptable methods of contraception include intrauterine device (IUD), oral contraceptive, subdermal implant and double barrier,
13. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
14. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 4.0),
15. Patients with a French social security in compliance with the Law relating to biomedical research (Article 1121-11 of French Public Health Code),
16. Voluntarily signed and dated written informed consent prior to any study specific procedure.

Exclusion Criteria:

1. Previous treatment with Trabectedin,
2. Currently active bacterial or fungus infection (> grade 2 CTC [CTCAE] HIV1, HIV2, hepatitis B or hepatitis C infections,
3. History of chronic alcohol use and/or cirrhosis,
4. The following unstable cardiac conditions are not allowed:

   * Congestive heart failure
   * Angina pectoris
   * Myocardial infarction within 1 year before registration
   * Uncontrolled arterial hypertension defined as blood pressure ≥ 150/100 mmHg despite optimal medical therapy
   * Arrhythmias clinically significant
5. Patients unable to receive corticotherapy,
6. Known central nervous system malignancy (CNS),
7. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding,
8. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
9. Previous enrolment in the present study,
10. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons,
11. Known hypersensitivity to any involved study drug or any of its formulation components.
12. Recent vaccination (in the last 2 weeks before inclusion) for yellow fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I (dose escalation sudy): 20 patients ; Phase II (interim analysis) : 16 patients ; Phase II (overall study): 30 patients.
Groups:
- Cohort 1: Trabectedin 0.30 mg/m2 IV + CP: Trabectedin 0.30 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 1 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 1: Trabectedin: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Patients will be allocated 4 doses of Trabectedin following a 3 + 3 design
  Phase 1: Cyclophosphamide: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
- Cohort 2: Trabectedin 0.40 mg/m2 IV + CP: Trabectedin 0.40 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 2 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 1: Trabectedin: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Patients will be allocated 4 doses of Trabectedin following a 3 + 3 design
  Phase 1: Cyclophosphamide: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
- Cohort 3: Trabectedin 0.50 mg/m2 IV + CP: Trabectedin 0.50 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 3 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 1: Trabectedin: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Patients will be allocated 4 doses of Trabectedin following a 3 + 3 design
  Phase 1: Cyclophosphamide: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
- Cohort 4: Trabectedin 0.60 mg/m2 IV + CP: Trabectedin 0.60 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 4 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 1: Trabectedin: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Patients will be allocated 4 doses of Trabectedin following a 3 + 3 design
  Phase 1: Cyclophosphamide: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
- Phase II: Trabectedin 0.50 mg/m2 IV + CP: Trabectedin 0.50 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in the phase II part of the study.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 2: Trabectedin: All patients will be treated at the RP2D of trabectedin defined in the preliminary phase I trial with the same schedule as in the phase I trial.
  Phase 2: Cyclophosphamide: All patients will be treated with metronomic cyclophosphamide with the same schedule as in the phase I trial.
Period: Phase I (Dose escalation part)
Arm/Group | Cohort 1: Trabectedin 0.30 mg/m2 IV + CP | Cohort 2: Trabectedin 0.40 mg/m2 IV + CP | Cohort 3: Trabectedin 0.50 mg/m2 IV + CP | Cohort 4: Trabectedin 0.60 mg/m2 IV + CP | Phase II: Trabectedin 0.50 mg/m2 IV + CP
Started | 3 | 3 | 7 | 7 | 0
Completed | 3 | 3 | 5 | 5 | 0
Not Completed | 0 | 0 | 2 | 2 | 0
Not completed — Clinical progression | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0
Period: Phase II
Arm/Group | Cohort 1: Trabectedin 0.30 mg/m2 IV + CP | Cohort 2: Trabectedin 0.40 mg/m2 IV + CP | Cohort 3: Trabectedin 0.50 mg/m2 IV + CP | Cohort 4: Trabectedin 0.60 mg/m2 IV + CP | Phase II: Trabectedin 0.50 mg/m2 IV + CP
Started | 0 | 0 | 0 | 0 | 30
Interim analysis (stage 2 of Simon's design) | 0 | 0 | 0 | 0 | 16
Completed | 0 | 0 | 0 | 0 | 24
Not Completed | 0 | 0 | 0 | 0 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Trabectedin 0.30 mg/m2 IV + CP: Trabectedin 0.30 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 1 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 1: Trabectedin: Phase I trial based on a dose escalating study design (3+3 traditional design) assessing four dose levels of Trabectedin in combination with metronomic cyclophosphamide (CP).
  A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.)
  Phase 1: Cyclophosphamide: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
- Cohort 2: Trabectedin 0.40 mg/m2 IV + CP: Trabectedin 0.40 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 2 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 1: Trabectedin: Phase I trial based on a dose escalating study design (3+3 traditional design) assessing four dose levels of Trabectedin in combination with metronomic cyclophosphamide (CP).
  A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.)
  Phase 1: Cyclophosphamide: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
- Cohort 3: Trabectedin 0.50 mg/m2 IV + CP: Trabectedin 0.50 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 3 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 1: Trabectedin: Phase I trial based on a dose escalating study design (3+3 traditional design) assessing four dose levels of Trabectedin in combination with metronomic cyclophosphamide (CP).
  A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.)
  Phase 1: Cyclophosphamide: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
- Cohort 4: Trabectedin 0.60 mg/m2 IV + CP: Trabectedin 0.60 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 4 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 1: Trabectedin: Phase I trial based on a dose escalating study design (3+3 traditional design) assessing four dose levels of Trabectedin in combination with metronomic cyclophosphamide (CP).
  A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.)
  Phase 1: Cyclophosphamide: A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
- Phase II: Trabectedin 0.50 mg/m2 IV + CP: Trabectedin 0.50 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in the phase II part of the study.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
  1 cycle = 28 days
  Phase 2: Trabectedin: Patients will be included in a single-arm phase II trial. Administrated dose will be the RP2D defined in the dose escalation part of the trial. The design will follow a two-stage Simon's optimal design.
  All patients will be treated at the RP2D of trabectedin defined in the preliminary phase I trial with the same schedule as in the phase I trial.
  Phase 2: Cyclophosphamide: All patients will be treated with metronomic cyclophosphamide with the same schedule as in the phase I trial.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Trabectedin 0.30 mg/m2 IV + CP | Cohort 2: Trabectedin 0.40 mg/m2 IV + CP | Cohort 3: Trabectedin 0.50 mg/m2 IV + CP | Cohort 4: Trabectedin 0.60 mg/m2 IV + CP | Phase II: Trabectedin 0.50 mg/m2 IV + CP | Total
Number analyzed (Participants) | 3 | 3 | 7 | 7 | 30 | 50
Age, Continuous [Median (Full Range); unit: years] | 61 [46 to 63] | 67 [50 to 73] | 61 [39 to 67] | 57 [27 to 69] | 67 [23 to 80] | 62.5 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 3 | 13 | 23
  Male | 1 | 0 | 5 | 4 | 17 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 7 | 7 | 30 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 3 | 3 | 7 | 7 | 30 | 50

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Trabectedin When Administered in Association With CP.
Description: MTD was determined by testing increasing doses of trabectedin up to 0.60 mg/m2 via IV on dose escalation cohorts 1 to 4 with 3 to 6 participants each.The MTD is defined as the highest dose at which no more than 1 in 6 of the patients in the cohort experienced a DLT in the first treatment cycle. See subsequent primary outcome measure for the DLT definition.
Time Frame: During the first cycle (28 days)
Population: 4 patients were not evaluable for MTD/DLT assessment.
Measure: Number; unit: mg/m^2
Groups:
- Phase I: Evaluable for Safety: All phase I patients received Trabectedin IV (3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks) in combination with CP (bi-daily (50 mg x 2) and given on a week on/week off ) according to the established dose escalation schedule. Patients who withdrew before completing the cycle 1 of treatment for other reason than DLT were not evaluable.
Arm/Group | Phase I: Evaluable for Safety
Number analyzed (Participants) | 16
mg/m^2 | 0.50

2. Primary Outcome: Phase I: Number of Patients Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as a treatment-related (at least possibly related) adverse event using the CTCAE V4.0, occuring during the fist cycle of treatment (28 days), that meets one of the following criteria:
  * Any grade-4 toxicity (except for vomiting without maximal symptomatic/prophylactic treatment)
  * Grade-3 non-haematological toxicity lasting > 7days (except for 1rst episode of nausea without maximal symptomatic/ prophylactic treatment and if toxicity is transaminitis, which may last > 7 days if total bilirubin is normal or grade-1)
  * Grade-3 hematologic toxicity lasting for > 7days
  * Grade 4 neutropenia with fever
  * Grade > 2 thrombocytopenia with bleeding
  * Is unrelated to disease, disease progression, inter-current illness, or concomitant medications.
Time Frame: During the first cycle (28 days)
Population: 4 patients were not evaluable for DLT evaluation as they did not complete the DLT assessment period: 2 in cohort 3 and 2 in cohort 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Trabectedin 0.30 mg/m2 IV + CP | Cohort 2: Trabectedin 0.40 mg/m2 IV + CP | Cohort 3: Trabectedin 0.50 mg/m2 IV + CP | Cohort 4: Trabectedin 0.60 mg/m2 IV + CP
Number analyzed (Participants) | 3 | 3 | 5 | 5
Participants | 0 | 0 | 0 | 2

3. Primary Outcome: Phase II: Percentage of Patients in Non-progression at 6 Months (RECIST V1.1)
Description: Non-progression is defined as complete or partial response (CR, PR) or stable disease (SD), as per RECIST v1.1. According to RECIST v1.1: Complete Response (CR) is defined as disappearance of all target lesions; Partial Response (PR) is defined as a >=30% decrease in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at baseline (SSD); Stable disease (SD) is defined as Neither sufficient shrinkage (compared to baseline) to qualify for PR or CR nor sufficient increase (taking as reference the SSD or while on study, whichever is smallest) to qualify for progressive disease (PD).
Time Frame: Phase II : 6 months after the start of treatment
Population: Stage 1 of Simon's design (interim analysis): 16 patients were included at this stage and 13 were evaluable for the primary endpoint.
  Stage 2 Simon's design (Final analysis): 30 patients were included at this stage and 24 were evaluable for the primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Trabectedin 0.50 mg/m2 IV + CP
Number analyzed (Participants) | 24
percentage of participants
  Interim analysis (Stage 1 of Simon's design): number analyzed (Participants) | 13
  Interim analysis (Stage 1 of Simon's design) | 23.1 [5.0 to 53.8]
  Overall (stage 2 of Simon's design) | 12.5 [2.7 to 32.4]

4. Secondary Outcome: Phase I: Percentage of Patients With Objective Response (RECIST V1.1)
Description: Objective response is defined as complete or partial response (CR, PR) as per RECIST v1.1. According to RECIST v1.1: Complete Response (CR) is defined as disappearance of all target lesions; Partial Response (PR) is defined as a >=30% decrease in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at baseline (SSD).
Time Frame: Throughout the treatment period, an average of 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 3: Trabectedin 0.50 mg/m2 IV + CP: Trabectedin 0.50 mg/m2 will be administered intravenously (IV), 3-hour infusion weekly for three consecutive weeks (days 1, 8 and 15) every 4 weeks, in cohort 3 of dose escalation.
  Cyclophosphamide (CP) will be administered bi-daily (50 mg x 2), and given on a week on/week off schedule.
Arm/Group | Cohort 1: Trabectedin 0.30 mg/m2 IV + CP | Cohort 2: Trabectedin 0.40 mg/m2 IV + CP | Cohort 3: Trabectedin 0.50 mg/m2 IV + CP | Cohort 4: Trabectedin 0.60 mg/m2 IV + CP
Number analyzed (Participants) | 3 | 3 | 5 | 5
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Phase II: Median Overall Survival
Description: Overall survival is defined as the time from the study initiation to death (any cause). Median overall survival was reported using kaplan-Meier method for calculation.
Time Frame: From start of treatment, and during treatment until death for any cause for up to 12 months.
Population: Stage 1 of Simon's design (interim analysis): 16 patients were included at this stage and 13 were evaluable for efficacy endpoints.
  Stage 2 Simon's design (Final analysis): 30 patients were included at this stage and 24 were evaluable for efficacy endpoints.
  The upper limit for the 95%CI for OS was not reached due to insufficient number of participants with events, and thus entered as "NA" (Not available).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Trabectedin 0.50 mg/m2 IV + CP
Number analyzed (Participants) | 24
months | 12.0 [5.8 to NA] — The upper limit for the 95%CI for OS was not reached due to insufficient number of participants with events, and thus entered as "NA" (Not available).

6. Secondary Outcome: Phase II: Median Profression-free Survival
Description: Progression-free survival is defined as the time from study treatment initiation to disease progression or death (of any cause), whichever occurs first. Progression is defined using RECIST v1.1, as a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), or a unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions. Median PFS was reported using kaplan-Meier method for calculation.
Time Frame: From start of treatment, and during treatment until progression or death for any cause for up to 12 months.
Population: Stage 1 of Simon's design (interim analysis): 16 patients were included at this stage and 13 were evaluable for efficacy endpoints.
  Stage 2 Simon's design (Final analysis): 30 patients were included at this stage and 24 were evaluable for efficacy endpoints.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Trabectedin 0.50 mg/m2 IV + CP
Number analyzed (Participants) | 24
months | 1.9 [1.7 to 4.4]

ADVERSE EVENTS:
Time Frame: Adverse events must be reported for 30 days after the last treatment administration or until the start of a new antitumor therapy, whichever occurs first. Phase I: approximatively 6 months after the start of study treatment. Phase II: approximatively 6 months after the start of study treatment.
Arm/Group | Cohort 1: Trabectedin 0.30 mg/m2 IV + CP | Cohort 2: Trabectedin 0.40 mg/m2 IV + CP | Cohort 3: Trabectedin 0.50 mg/m2 IV + CP | Cohort 4: Trabectedin 0.60 mg/m2 IV + CP | Phase II: Trabectedin 0.50 mg/m2 IV + CP
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 4/5 | 4/5 | 20/30
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/5 | 2/5 | 20/30
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5 | 5/5 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Trabectedin 0.30 mg/m2 IV + CP (N=3) | Cohort 2: Trabectedin 0.40 mg/m2 IV + CP (N=3) | Cohort 3: Trabectedin 0.50 mg/m2 IV + CP (N=5) | Cohort 4: Trabectedin 0.60 mg/m2 IV + CP (N=5) | Phase II: Trabectedin 0.50 mg/m2 IV + CP (N=30)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 4 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening of GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestine obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema lower limb (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decompensation cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cruralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vein compression (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exeresis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Trabectedin 0.30 mg/m2 IV + CP (N=3) | Cohort 2: Trabectedin 0.40 mg/m2 IV + CP (N=3) | Cohort 3: Trabectedin 0.50 mg/m2 IV + CP (N=5) | Cohort 4: Trabectedin 0.60 mg/m2 IV + CP (N=5) | Phase II: Trabectedin 0.50 mg/m2 IV + CP (N=30)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 19 (21)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 11 (13)
Diarrhea (Gastrointestinal disorders) | 2 (6) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Aphta (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Black stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food disgust (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 8 (8)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 4 (6) | 4 (8) | 20 (26)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 15 (17)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Edema limbs (General disorders) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 6 (6)
Fatigue (General disorders) | 3 (4) | 3 (3) | 2 (2) | 5 (6) | 27 (32)
Fever (General disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 4 (5)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac Chest pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site condition - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ankle sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 12 (14)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 10 (10)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 6 (9)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
GGT increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 8 (8)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 26 (26)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 11 (13)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 7 (11)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
LDH increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperleukocytosis (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermittent monocytosis (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 9 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ante-brachial flexion restriction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vesicular murmur diminution (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythemato-vesicular eruption (zona type (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT02805725/Prot_SAP_000.pdf